CLINICAL TRIAL: NCT03652220
Title: Meditation Based Lifestyle Modification in Depression: a Randomized Controlled Trial
Brief Title: Meditation Based Lifestyle Modification in Depression
Acronym: MBLM-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonie Kliniken Zschadraß (Other)
Collaborators: Charite University, Berlin, Germany (Other); Chemnitz University of Technology (Other)
Responsible Party: Principal Investigator, Holger C. Bringmann, Dr. med. B. Sc., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBLM-D
Record Dates: First submitted 2018-08-22; First posted 2018-08-29 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Intervention Model Description: This is a three-arm, randomized, active-controlled, unblinded, parallel, exploratory study to compare the outcome in depression between standard specific treatment, multimodal specific treatment and standard treatment plus MBLM. After being screened for eligibility and signing the informed consent patients will be randomized 1:1:1 to either one of the groups. After being enrolled, patients in MBLM group receive an introductory education of the MBLM course and then join group sessions weekly for 8 weeks. They also see a consultant psychiatrist as needed for drug continuation therapy. Patients should practice MBLM related content at home for a proposed duration of 30-45 minutes per day. Patients in the control groups receive standard (control group I) or multimodal (control group II) treatment as administered by their consultant psychiatrist.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): 8 weeks Minimal treatment + MBLM 16 weeks Multimodal specific treatment + MBLM Consolidation
  Definitions Minimal treatment: drug continuation under medical supervision Multimodal specific treatment: Drugs / Psychotherapy / Excercise therapy / Ergotherapy / Relaxation; excl. Yoga, Mantra, MBSR MBLM: 8-week course Meditation Based Lifestyle Modification MBLM-Consolidation: weekly Mantra-Meditation, monthly Life-Ethics
  Interventions: Behavioral: Meditation Based Lifestyle Modification
- Control I (Active Comparator): 8 weeks Minimal treatment 16 weeks Multimodal specific treatment
  Definitions Minimal treatment: drug continuation under medical supervision Multimodal specific treatment: Drugs / Psychotherapy / Excercise therapy / Ergotherapy / Relaxation; excl. Yoga, Mantra, MBSR MBLM: 8-week course Meditation Based Lifestyle Modification MBLM-Consolidation: weekly Mantra-Meditation, monthly Life-Ethics
  Interventions: Other: Minimal treatment; Other: Multimodal specific treatment:
- Control 2 (Active Comparator): Definitions 24 weeks Multimodal specific treatment
  Minimal treatment: drug continuation under medical supervision Multimodal specific treatment: Drugs / Psychotherapy / Excercise therapy / Ergotherapy / Relaxation; excl. Yoga, Mantra, MBSR MBLM: 8-week course Meditation Based Lifestyle Modification MBLM-Consolidation: weekly Mantra-Meditation, monthly Life-Ethics
  Interventions: Other: Multimodal specific treatment:

INTERVENTIONS:
Behavioral: Meditation Based Lifestyle Modification — 8 weekly modules, each 3.5 hours of Life ethics, Yoga exercises and Mantra Meditation
  Arms: Intervention
Other: Minimal treatment — Drug continuation under medical supervision
  Arms: Control I
Other: Multimodal specific treatment: — Drugs / Psychotherapy / Excercise therapy / Ergotherapy / Relaxation; excl. Yoga, Mantra, MBSR
  Arms: Control 2; Control I

SUMMARY:
To evaluate effectiveness of a 8-week behavioral Mind-Body-Intervention based on Yoga and Meditation in depressive outpatients.

DETAILED DESCRIPTION:
As a contribution to the field of Integral Medicine, Meditation Based Lifestyle Modification (MBLM) is a holistic therapy for patients with mental disorders. Influenced by Ayurveda and Yoga, it uses mantra meditation, ethical conduct and healthy life style to promote physical, mental and spiritual health. MBLM explains processes within the body and the mind and their relation to diet, exercise, biorhythms, social and personal conduct in an easy but profound way and on an experiential level. Besides providing tools for physical, mental and emotional self-regulation, MBLM lays ground for personal growth and transcendence of the mind. It is intended to be implemented in groups of patients as well as individual daily training, and because of its modular structure can be adjusted in intensity, duration and weighting of the components according to the specific needs and disorders to be addressed. This makes it also eligible for its potential use in prevention of mental disease and treatment of psychic comorbidities in patients with chronic somatic illness.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria to be enrolled:

1. Outpatients
2. Written informed consent by patients who are competent to consent to study participation
3. Diagnosis of current mild or moderate episode of depression diagnosed by a consultant psychiatrist
4. Male or female ≥18 years of age
5. BDI-II >= 10
6. Patients must be physically able to perform simple Yoga postures and to sit silently for 20 minutes

Exclusion Criteria:

Patients will be excluded for ANY ONE of the following reasons:

1. Psychotic Symptoms
2. Acute suicidal tendencies
3. Compulsive disorders
4. Cerebro-organic diseases with clinically relevant symptoms
5. Severe multimorbidity
6. Clinically relevant addictions (tobacco abuse or addiction is allowed)
7. Current participation in another trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Change of Beck Depression Index BDI-II | Baseline, 4 weeks, 8 weeks. Follow-up 24 weeks
  Change of depressive Symptoms

SECONDARY OUTCOMES:
Freiburg Mindfulness Inventory (FMI) | Baseline, 8 weeks; Follow-up 24 weeks
  The FMI (14 item version; FMI-14) is a widely used instrument that assesses trait mindfulness that has been validated in a number of studies. This short form of the originally 30-items questionnaire provides robust and psychometrically stable (alpha = .86) properties. It is semantically independent from a Buddhist or meditation context (Walach, Buchheld, Buttenmüller, Kleinknecht, & Schmidt, 2006).
Mindful Attention Awareness Scale (MAAS) | Baseline, 8 weeks; Follow-up 24 weeks
  The MAAS (K. W. Brown & Ryan, 2003) is a 15-item scale designed to assess a core characteristic of dispositional mindfulness, namely, open or receptive awareness of and attention to what is taking place in the present. The scale shows strong psychometric properties and has been validated with college, community, and cancer patient samples. Correlational, quasi-experimental, and laboratory studies have shown that the MAAS taps a unique quality of consciousness that is related to, and predictive of, a variety of self-regulation and well-being constructs.
Perceived Stress Scale (PSS-10) | Baseline, 8 weeks; Follow-up 24 weeks
  The Perceived Stress Scale (Cohen, Kamarck, & Mermelstein, 1983) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes a number of direct queries about current levels of experienced stress.
Brief Symptom Checklist (BSI-18) | Baseline, 8 weeks; Follow-up 24 weeks
  The BSI-18 (Franke et al., 2017) contains the three six-item scales somatization, depression, and anxiety as well as the Global Severity Index (GSI), including all 18 items. The BSI-18 is the latest and shortest of the multidimensional versions of the commonly used Symptom-Checklist 90-R.
Aachen Self-Efficacy Questionnaire (Aachener Selbstwirksamkeitsfragebogen, [ASF]) | Baseline, 8 weeks; Follow-up 24 weeks
  The ASF assesses generalized self-efficacy as well as specific factors such as achievement, social interaction and body- related self esteem. Its internal consistency (Chronbach's α) is 0.90 for the general scale, and 0.74-0.84 for its subscales. The test-retest reliability for the ASF is rtt 0.66 over a period of eight weeks (Flatten, Wälte, & Perlitz, 2008).
SpREUK-P-SF17 | Baseline, 8 weeks; Follow-up 24 weeks
  This instrument (Bussing, Reiser, Michalsen, & Baumann, 2012) was designed to measure the engagement frequencies of a large spectrum of organized and private religious, spiritual, existential and philosophical practices. It avoids the intermix of cognitive / emotional attitudes and convictions on the one hand with the engagement in forms of practice (action, behaviour) on the other. To account for the fact of institutional religiosity declines not only in Europe, and the alternative use of various existing esoteric and religious resources, the instrument differentiates both the frequency of conventional forms of spirituality/religiosity, and also more reflecting or philosophical practice and nature/environment- oriented practices.
Triguna Scale (TGS) | Baseline, 8 weeks; Follow-up 24 weeks
  TGS is an instrument to rate a variety of psychosocial traits (e.g. cognition, motivation, social behavior etc.) according to tri-guna model of Yoga philosophy (M. Puta, 2016; Maika Puta & Sedlmeier, 2014). The reliability of the majority of the 27 scales corresponds to reliability values of established personality inventories: Cronbach's α of 24 subscales is above .7. The internal consistencies of the other three subscales don't meet this standard, but their values are still above .6. Measures determining the validity of the inventory are very good. The exploratory factor analysis of the second study shows that all scales consist of three factors, each of which can be related to one of the gunas.
Transgression-Related Interpersonal Motivations Inventory (TRIM) | Baseline, 8 weeks; Follow-up 24 weeks
  The TRIM is a self-report instrument that assesses the motivations assumed to underlie forgiving: Avoidance and Revenge. Responses to 12 statements referring to a transgression recipient's current thoughts and feelings about the transgressor are scored on a 5-point Likert-type scale. Recently, a six-item subscale to reflect benevolent motivations toward the transgressor has been under development (contact the first author for details). The TRIM subscales not only correlate with a variety of relationship, offense, and social-cognitive variables, they have also demonstrated strong relationships to a single-item measure of forgiveness. The inventory takes approximately 5 minutes to complete (McCullough et al., 1998).
Brief global measure of client satisfaction (ZUF-8) | Baseline, 8 weeks; Follow-up 24 weeks
  ZUF-8 is a global, one-dimensional patient satisfaction measurement tool. It is the German-language adaptation of the American CSQ-8 by Attkisson & Zwick (1982). Over eight items, the general satisfaction with aspects of the clinic or the received treatment is recorded. ZUF-8 is particularly suitable for economical screening of patient satisfaction (Schmidt, Lamprecht, & Wittmann, 1989).
Perseverative Thinking Questionnaire (PTQ) | Baseline, 8 weeks; Follow-up 24 weeks
  The PTQ (Ehring et al., 2011) is a 15-item questionnaire assessing the tendency to engage in repetitive negative thinking independent of a disorder-specific content. Items are rated on a scale ranging from 0 (never) to 4 (almost always). The PTQ consists of three subscales: Core features of repetitive negative thinking (sample item: 'The same thoughts keep going through my mind again and again'.), perceived unproductiveness of repetitive negative thinking (sample item: 'I keep asking myself questions without finding an answer'.), and repetitive negative thinking capturing mental capacity (sample item: 'My thoughts prevent me from focusing on other things'.). Confirmatory factor analysis provides support for a 3-factor solution.
Duke University Religion Index (DUREL) | Baseline, 8 weeks; Follow-up 24 weeks
  The Duke University Religion Index (DUREL) is a five-item measure of religious involvement, and was developed for use in large cross-sectional and longitudinal observational studies. The instrument assesses the three major dimensions of religiosity that were identified during a consensus meeting sponsored by the National Institute on Aging. Those three dimensions are organizational religious activity, non-organizational religious activity, and intrinsic religiosity (or subjective religiosity). The DUREL measures each of these dimensions by a separate "subscale", and correlations with health outcomes should be analyzed by subscale in separate models.
Aspects of Spirituality (ASP) | Baseline, 8 weeks; Follow-up 24 weeks
  The ASP questionnaire was developed to measure a wide variety of vital aspects of spirituality beyond conventional conceptual boundaries in secular societies. Both expert representatives of various spiritual orientations and also atheists were asked which aspects of spirituality are relevant to them (Büssing, 2006). Identified motifs we condensed to 40 items of the Aspects of Spirituality (ASP 1.0) questionnaire (7 factors; Cronbach ́s alpha = .94) (Büssing et al., 2007) which differentiates and quantifies cognitive, emotional, intentional and action-oriented matters of theism/belief, (esoteric) transcendence, existentialism, humanism etc. The reliable and valid instrument is suited to be used in health care research (Büssing et al. 2007).
Spirituality as a Resource to Rely on in Chronic Illness (SpREUK-15) | Baseline, 8 weeks; Follow-up 24 weeks
  The SpREUK was developed to investigate whether or not patients with chronic diseases living in secular societies rely on spirituality as a resource to cope with illness. The SpREUK questionnaire relies on essential motifs found in counseling interviews with chronic disease patients (i.e., having trust/faith; search for a transcendent source to rely on; reflection of life and subsequent change of life and behavior). The instrument is suited to be used in health care research (A Büssing, Ostermann, & Matthiessen, 2005).
Assessment of training and exercise hours | Daily for 8 weeks in intervention group
  Patients receive weekly working sheets to document daily, cumulative duration of practice.
Heart Rate Variability | 24h continuous measurement at Baseline, and at 8 weeks
  Faros eMotion 180 derived 3-lead ECG Heart Rate Variability (RR-Intervals in ms)
Heart Rate | 8 weeks continuously in 1-minute intervals
  FitBit Charge 2 derived Heart Rate (beats per minute)
Sleep duration | 8 weeks continuously
  FitBit Charge 2 derived sleep duration in minutes
Activity: Steps per day | 8 weeks continuously
  FitBit Charge 2 derived steps per day
Qualitative Interview | After 8 or 24 weeks
  A single qualitative interview with selected patients (around 10 patients in each group) will be held after at least 8 weeks of treatment to assess qualitative data:
  Interviews will involve the following domains of exploration
  1. How has the treatment you have received during the last weeks has affected your depression?
  2. How did you experience the treatment?
  3. What does spirituality mean to you and how has that changed during the treatment?
  Interviews are an optional part of the study in terms of a mixed model approach to receive quantitative and qualitative data as well. Participants willing to be interviewed have to sign an additional consent for the collection and processing of personal interview data.

CONTACTS AND LOCATIONS:
Locations (1):
- Diakoniekliniken Zschadraß, Colditz, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bringmann HC, Berghofer A, Jeitler M, Michalsen A, Brunnhuber S, Haller H. Meditation-Based Lifestyle Modification in Mild-to-Moderate Depression: Outcomes and Moderation Effects of Spirituality. J Integr Complement Med. 2024 Jun;30(6):532-542. doi: 10.1089/jicm.2023.0179. Epub 2023 Nov 27. PMID 38011739
- [Derived] Bringmann HC, Vennemann J, Gross J, Matko K, Sedlmeier P. "To Be Finally at Peace with Myself": A Qualitative Study Reflecting Experiences of the Meditation-Based Lifestyle Modification Program in Mild-to-Moderate Depression. J Altern Complement Med. 2021 Sep;27(9):786-795. doi: 10.1089/acm.2021.0038. Epub 2021 Jun 29. PMID 34185550